CLINICAL TRIAL: NCT01093183
Title: A Phase I/II Clinical Trial of Lenalidomide in Combination With Oral Cyclophosphamide in Patients With Previously Treated Hormone Refractory Prostate Cancer
Brief Title: Lenalidomide and Cyclophosphamide in Treating Patients With Previously Treated Hormone-Refractory Prostate Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: study sponsors withdrew support for the study drug.
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0479-09-FB; NCI-2010-00363 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 479-09 (Other: University of Nebraska Medical Center); P30CA036727 (NIH)
Record Dates: First submitted 2010-03-24; First posted 2010-03-25 (Estimated); Results first posted 2018-06-11 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Adenocarcinoma of the Prostate; Hormone-resistant Prostate Cancer; Recurrent Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Lenalidomide; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (lenalidomide and cyclophosphamide) (Experimental): Patients receive lenalidomide PO QD on days 1-21 and cyclophosphamide PO QD on days 1-28. Treatment repeats every 28 days for at least 4 courses in the absence of disease progression or unacceptable toxicity. Treatment modifications may apply according to response.
  Interventions: Drug: lenalidomide; Drug: cyclophosphamide; Other: laboratory biomarker analysis; Other: questionnaire administration; Other: quality-of-life assessment

INTERVENTIONS:
Drug: lenalidomide — Given PO
  Other Names: CC-5013; IMiD-1; Revlimid
Drug: cyclophosphamide — Given PO
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Other: laboratory biomarker analysis — Correlative studies
Other: questionnaire administration — Ancillary studies
Other: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
This phase I/II trial studies the side effects and best dose of lenalidomide when given together with cyclophosphamide and to see how well they work in treating patients with previously treated hormone-refractory prostate cancer. Lenalidomide may stop the growth of prostate cancer by blocking blood flow to the tumor. Drugs used in chemotherapy, such as cyclophosphamide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving lenalidomide together with cyclophosphamide may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) and the dose limiting toxicities (DLT) of lenalidomide administered in combination with oral cyclophosphamide.

SECONDARY OBJECTIVES:

I. To evaluate the objective prostate-specific antigen (PSA) response (50% decrease in PSA levels sustained for at least 4 weeks) as defined by PSA working group criteria; or a decrease in absolute PSA or a decrease in PSA velocity, increase in PSA doubling time, duration of any responses.

II. To explore the anti-tumor activity of the combination of lenalidomide plus oral cyclophosphamide in patients with previously treated hormone refractory prostate cancer.

III. To evaluate baseline and change of quality of life, particularly, bone pain and analgesic consumption, of the patients on this combination chemotherapy.

TERTIARY OBJECTIVES:

I. To determine whether related cytokines and biomarkers (serum levels of tumor necrosis factor-alpha, basic fibroblast growth factor, vascular endothelial growth factor [VEGF], T cell inhibitory activity, phytohemagglutinin [PHA] and interleukin [IL]-2, mononuclear cell isolation, VEGF, basic fibroblast growth factor [bFGF], IL-6) can help predict response to patients undergoing treatment with lenalidomide and cyclophosphamide.

OUTLINE: This is a phase I, dose-escalation study of lenalidomide followed by a phase II study.

Patients receive lenalidomide orally (PO) once daily (QD) on days 1-21 and cyclophosphamide PO QD on days 1-28. Treatment repeats every 28 days for at least 4 courses in the absence of disease progression or unacceptable toxicity. Treatment modifications may apply according to response.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status of 2 or less
* Men with histologically documented previously treated hormone refractory adenocarcinoma of the prostate; mixed histology and rare subtypes histology of prostate cancer are allowed only in phase 1 portion of trial
* Patients must be on an luteinizing-hormone-releasing hormone (LHRH) agonist or have undergone surgical castration
* Patients must have already failed or progressed after treatment with a docetaxel-based regimen; patients who were unable to tolerate docetaxel are eligible in phase 1 portion of trial
* Creatinine clearance >= 45 by Cockcroft-Gault formula
* Total bilirubin =< upper limit of normal (ULN)
* Aspartate aminotransferase (AST) < 2 x ULN
* Alanine aminotransferase (ALT) < 2 x ULN
* Hepatic alkaline phosphatase < 2 x ULN (< 5.0 x ULN for subjects with known bone metastases)
* Absolute neutrophil count greater than 1,500/mm^3
* Platelets greater than 100,000/mm^3
* Hemoglobin >= 9.0 g/dL
* Able to adhere to the study visit schedule and other protocol requirements
* No serious disease or condition that, in the opinion of the investigator, would compromise the patient's ability to participate in the study
* All study participants must be registered into the mandatory Revlimid REMS program, and be willing and able to comply with the requirements of Revlimid REMS
* Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to acetylsalicylic acid [ASA] may use warfarin or low molecular weight heparin)
* Men must agree to use a latex condom during sexual contact with females of childbearing potential (FCBP) even if they have had a successful vasectomy
* Male subject agrees to use an acceptable method for contraception for the duration of the study
* Electrocardiogram (EKG) at baseline, if abnormal, not medically relevant

Exclusion Criteria:

* Treatment with a cytotoxic chemotherapy or investigational drug within 30 days before day 1 of study treatment; palliative radiation therapy is allowed, as long as a radiated lesion is not used to assess response rate, and the radiation occurred greater than 4 weeks prior to enrollment
* Known positive for human immunodeficiency virus (HIV) or infectious hepatitis, type A, B or C or active hepatitis
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form
* Known hypersensitivity to thalidomide, lenalidomide or cyclophosphamide
* Active infection at the start of lenalidomide
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities; prior to study entry, any EKG abnormality at screening has to be documented by the investigator as not medically relevant
* History of life threatening or recurrent thrombosis/embolism; patients may participate if they are adequately anti-coagulated during the treatment
* Patient has > grade 2 peripheral neuropathy within 14 days before enrollment
* Any evidence of severe or uncontrolled systemic disease (e.g., unstable or uncompensated respiratory, cardiac, hepatic, or renal disease)
* Any unresolved chronic toxicity greater than Common Terminology Criteria (CTC) grade 2 from previous anticancer therapy (except alopecia)
* Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the subject to participate in the trial

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-03-04 (Actual); Primary Completion 2015-05-19 (Actual); Study Completion 2015-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James K Schwarz, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I Treatment (Lenalidomide and Cyclophosphamide); Phase II Treatment (Lenalidomide and Cyclophosphamide): Patients receive lenalidomide PO QD on days 1-21 and cyclophosphamide PO QD on days 1-28. Treatment repeats every 28 days for at least 4 courses in the absence of disease progression or unacceptable toxicity. Treatment modifications may apply according to response.
  lenalidomide and cyclophosphamide: Given PO
Period: Overall Study
Arm/Group | Phase I Treatment (Lenalidomide and Cyclophosphamide) | Phase II Treatment (Lenalidomide and Cyclophosphamide)
Started | 19 | 6
Completed | 18 | 4
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Population: 19 patients were treated on the dose-escalation phase I, and an additional 6 patients received treatment in the expansion phase II.
Groups:
- Treatment (Lenalidomide and Cyclophosphamide): Patients receive lenalidomide PO QD on days 1-21 and cyclophosphamide PO QD on days 1-28. Treatment repeats every 28 days for at least 4 courses in the absence of disease progression or unacceptable toxicity. Treatment modifications may apply according to response.
  lenalidomide and cyclophosphamide: Given PO
Arm/Group | Treatment (Lenalidomide and Cyclophosphamide)
Number analyzed (Participants) | 25
Age, Continuous [Median (Full Range); unit: years] | 76 [50 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 25
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Lenalidomide Administered in Combination With Oral Cyclophosphamide (Phase I)
Description: Defined to be the dose cohort below which 2 of 3 or 3 of 6 patients experience dose-limiting toxicities in course 1 or the highest dose cohort of 25 mg.
Time Frame: 28 days
Measure: Number; unit: mg
Arm/Group | Treatment (Lenalidomide and Cyclophosphamide)
Number analyzed (Participants) | 19
mg | 25

2. Secondary Outcome: Number of Patients Achieving Objective PSA Response (50% Decrease in PSA Levels Sustained for at Least 4 Weeks) as Defined by PSA Working Group Criteria
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Lenalidomide and Cyclophosphamide)
Number analyzed (Participants) | 22
Participants | 7

3. Secondary Outcome: Anti-tumor Activity as Assessed by the Sum of Complete Response (CR), Partial Response (PR), and Stable Disease (SD)
Description: As measured by Response Evaluation Criteria In Solid Tumors (RECIST version 1.1), in which CR is defined as disappearance of target lesions and a partial response (PR) is defined as at least a 30% decrease in the sum of the longest diameter of target lesions. PD is defined as 20% increase over smallest sum on study (including baseline if that is smallest) and at least 5 mm increase or new lesions. SD is defined as not enough response to be PR and not enough progression to be PD.
Time Frame: Up to 4 months
Population: Of the 22 subjects evaluable, three patients did not complete 2 cycles of therapy to reassess or response evaluation.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Lenalidomide and Cyclophosphamide)
Number analyzed (Participants) | 22
Participants
  Stable disease | 15
  partial response | 7

4. Secondary Outcome: Proportion of Patients Achieving CR
Time Frame: At 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Lenalidomide and Cyclophosphamide)
Number analyzed (Participants) | 22
Participants | 0

5. Secondary Outcome: Overall Survival
Time Frame: Up to 4 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Lenalidomide and Cyclophosphamide)
Number analyzed (Participants) | 25
months | 20 [13 to 24]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time the first patient enrolled through when the last patient completed study treatment.
Arm/Group | Treatment (Lenalidomide and Cyclophosphamide)
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 6/25
Other Adverse Events (participants affected / at risk) | 20/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Lenalidomide and Cyclophosphamide) (N=25)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) — low white blood cell count
Neutropenia (Blood and lymphatic system disorders) | 2 (2) — low neutrophil cell count
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) — low platelet cell counts
Hypotension (Vascular disorders) | 1 (1) — a blood pressure that is below the normal expected for an individual
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Vasovagal episode (Nervous system disorders) | 1 (1)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (2) — a reduction in the amount of hemoglobin in 100 ml of blood.
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1) — an ANC <1000/mm3 and a single temperature of >38.3 degrees C (101 degrees F) or a sustained temperature of >=38 degrees C (100.4 degrees F) for more than one hour.
Lung Infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Lenalidomide and Cyclophosphamide) (N=25)
Fatigue (General disorders) | 4 (4)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) — laboratory test results that indicate a low concentration of potassium in the blood
Neutropenia (Blood and lymphatic system disorders) | 6 (13)
Leukopenia (Blood and lymphatic system disorders) | 4 (9) — low white blood cell counts
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2) — laboratory test results that indicate a low concentration of phosphates in the blood
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (5)
Alkaline Phosphatase Increased (Investigations) | 2 (2) — laboratory test results that indicate an increase in the level of alkaline phosphatase in a blood specimen

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No